CLINICAL TRIAL: NCT06726161
Title: Phase 1/1b Single Arm, Open-label Trial of Theranostic Pair RYZ811 (Diagnostic) and RYZ801 (Therapeutic) to Identify and Treat Subjects With GPC3+ Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Study of the Theranostic Pair RYZ811 (Diagnostic) and RYZ801 (Therapeutic) to Identify and Treat Subjects With GPC3+ Unresectable HCC
Acronym: GPC3
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RayzeBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RYZ801-101
Record Dates: First submitted 2024-11-05; First posted 2024-12-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: HCC
Keywords: actinium; theranostic; alpha-emitter; RYZ811; RYZ801; 225Ac; HCC; targeted radiotherapy; radiopharmaceutical; unresectable HCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation, Dose Expansion (Experimental)
  Interventions: Diagnostic Test: RYZ811; Drug: RYZ801

INTERVENTIONS:
Diagnostic Test: RYZ811 — Ga-68
Drug: RYZ801 — Ac-225

SUMMARY:
A single arm, open-label Phase 1/1b study of the theranostic pair RYZ811 (diagnostic) and RYZ801 (therapeutic) to identify and treat subjects with GPC3+ unresectable HCC

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years at the time of signing the informed consent form (ICF)
* Histologically/cytologically confirmed diagnosis of HCC.
* Barcelona Clinic Liver Cancer (BCLC) Stage C or BCLC Stage B not amenable to locoregional therapy
* Child-Pugh A
* ECOG PS 0-1
* At least 1 prior systemic therapy for unresectable HCC
* Measurable disease per RECIST v1.1
* Sufficient renal function
* Adequate hematologic function
* Adequate hepatic function
* The subject must have recovered from toxicities related to prior treatments to ≤Grade 1, unless clinically nonsignificant and/or stable on supportive therapy
* If HBV or HCV infection: Disease managed per local practice; antiviral treatment is allowed.
* Gastric or esophageal varices previously treated with endoscopic therapy according to institutional standards are permitted if no clinically significant bleeding
* For women of childbearing potential (WOCBP):

  * Negative serum pregnancy test within 48 hours prior to the first dose of RYZ811
  * Agreement to use barrier contraception and a second form of highly effective contraception
* For sexually active males:

  * Must use a condom during intercourse
  * Male subjects whose sexual partners are WOCBP must also agree to use a second form of highly effective contraception
  * A condom is required to be used also by vasectomized men

Exclusion Criteria:

* Subjects with fibrolamellar carcinoma, sarcomatoid HCC or combined hepatocellular cholangiocarcinoma
* Prior liver transplantation or candidates for liver transplantation
* Known hypersensitivity to 68Ga, 225Ac or any of the excipients of RYZ811 or RYZ801
* Portal vein tumor thrombosis classified as Vp4
* Documented hepatic encephalopathy
* Clinically meaningful ascites
* Prior EBRT to the liver
* Prior EBRT to >25% of the bone marrow
* Prior liver radioembolization
* Previously treated central nervous system (CNS) metastasis without recovery from acute side effects
* Documented history of idiopathic pulmonary fibrosis (IPF), interstitial lung disease (ILD) or pneumonitis
* Uncontrolled significant intercurrent illness including, but not limited to:

  * QT interval corrected for heart rate using Fridericia's formula (QTcF) >470 ms
  * Hemoglobin A1c (HgB A1c) ≥8%
  * Uncontrolled hypertension
  * Significant cardiovascular disease or heart failure
* History of clinically significant bleeding
* Prior participation in any interventional clinical study
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study
* Have a history of primary malignancy within the past 3 years other than (1) HCC, (2) adequately treated carcinoma in situ or non-melanoma carcinoma of the skin, (3) any other curatively treated malignancy that is not expected to require treatment for recurrence during participation in the study, or (4) an untreated cancer on active surveillance that may not affect the subject's survival status for >3 years
* Subject requires other treatment that in the opinion of the Investigator would be more appropriate than what is offered in the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic - RYZ801 | Rate of DLTs during the first 42 days of study treatment
  To determine the RP2D of RYZ801 in subjects with GPC3+ unresectable HCC (Dose Escalation only)
Therapeutic - RYZ801 | Baseline, before and after each RYZ801 treatment cycle. For the Dose Escalation, Cycle 1 is 42 days. All other cycles are 28 days.
  To assess the safety and tolerability of RYZ801 in subjects with GPC3+ unresectable HCC. Safety and tolerability of RYZ801 as measured by incidence and severity of AEs, including SAEs, laboratory changes, and other safety findings.
Diagnostic - RYZ811 | Baseline, pre-injection and post-injection (up to 144 hours post RYZ811 injection).
  To assess the safety and tolerability of RYZ811 in subjects with unresectable HCC. Safety and tolerability of RYZ811 as measured by incidence and severity of AEs, including SAEs, laboratory changes, and other safety findings.
Diagnostic - RYZ811 | RYZ811 biodistribution to be assessed by PET/CT at 1, 2 and 3 hours post-injection.
  To evaluate the biodistribution of RYZ811 in subjects with unresectable HCC. SUV (mean, maximum and peak) of organs and tumors; volume of RYZ811 avid uptake in tumor lesions; and tumor-to-normal organ tracer uptake ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Heying Duan, MD, Study Director — RayzeBio, Inc.
Locations (2):
- United States (2):
  - Research Facility, Birmingham, Alabama
  - Research Facility, Grand Rapids, Michigan